CLINICAL TRIAL: NCT02002312
Title: Phase II Study Of Lutetium-177 Labeled Chimeric Monoclonal Antibody Girentuximab (177Lu-DOTA-girentuximab) in Patients With Advanced Renal Cell Cancer
Brief Title: Phase II Study of Lutetium-177 Labeled Girentuximab in Patients With Advanced Renal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO2009/322
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
Keywords: Advanced Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma (ccRCC); Lutetium-177; Lu-177; girentuximab; cG250; Monoclonal Antibody
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lu-177-DOTA-girentuximab (Experimental): Patients in receive 10 mg of girentuximab coupled to DOTA and labeled with 65 mCi/m2 of Lu-177 if targeting of In-111-DOTA-girentuximab is observed in at least 1 lesion. Patients may be retreated no sooner than 12 weeks after the prior treatment with a dose of no more than 75% of the previous dose, for a total of not more than three treatments.
  Interventions: Drug: Lu-177-DOTA-girentuximab

INTERVENTIONS:
Drug: Lu-177-DOTA-girentuximab — Drug: In-111-DOTA-girentuximab At day 1, every patient received girentuximab at a dose of 10 mg coupled to DOTA and labeled with 5 mCi of In-111.
  Drug: Lu-177-DOTA-girentuximab At day 8-10, every patient receives girentuximab at a dose of 10 mg coupled to DOTA and labeled with 65 mCi/m2 of Lu-177. If eligible, patients are retreated at a dose 75% of the previous dose, for a total of not more than three treatments.
  Other Names: Lu-177-DOTA-cG250

SUMMARY:
To determine the efficacy of multiple doses Lutetium-177-DOTA-girentuximab in patients with advanced clear cell renal cell carcinoma using RECIST criteria.

DETAILED DESCRIPTION:
This is a Phase II study using Lu-177-DOTA-girentuximab for treatment of patients with advanced clear cell renal cell carcinoma. The trial requires 14 patients. CT scans will be carried out at baseline and after 12 weeks, for response assessment using RECIST criteria.

Patients will initially receive 5 mCi/10 mg Indium-111-DOTA-girentuximab antibody (an imaging dose preceeding Lu-177-girentuximab treatment). Whole body and blood measurements of radioactivity will be obtained on at least three occasions for one week to determine targeting and dosimetry. Only if at least one known and evaluable metastatic lesion is visualized with In-111-DOTA-girentuximab, therapeutic Lu-177-DOTA- girentuximab will be administered the following week. In the absence of disease progression and after recovery from toxicity, patients may be retreated no sooner than 12 weeks after the prior treatment with a dose of no more than 75% of the previous dose, for a total of not more than three treatments. Only patients who have normal pharmacokinetics on the preceding diagnostic In-111-girentuximab study (indicative of human antichimeric antibodies (HACA) negativity) are eligible for retreatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with proven advanced and progressive RCC of the clear cell type
* Presence of RECIST v.1.1 evaluable lesions, all < 5 cm
* Performance status: Karnofsky > 70 %
* Laboratory values: • White blood cells (WBC) > 3.5 x 109/l • Platelet count > 150 x 109/l • Hemoglobin > 6 mmol/l • Total bilirubin < 2 x upper limit of normal (ULN) • ASAT, ALAT < 3 x ULN (< 5 x ULN if liver metastases present) • MDRD ≥ 40 ml/min
* Negative pregnancy test for women of childbearing potential (urine or serum)
* Age over 18 years
* Written informed consent

Exclusion criteria:

* Known or suspected CNS metastases including leptomeningeal metastases. History or clinical evidence of (CNS) metastases (unless they are previously-treated CNS metastases and patients meet all 3 of the following criteria: are asymptomatic, have had no evidence of active CNS metastases for ≥3 months prior to enrollment, and have had no requirement for steroids or enzyme inducing anticonvulsants in the last 14 days)
* Untreated hypercalcemia
* Chemotherapy, external beam radiation, immunotherapy or angiogenesis inhibitors or mTOR inhibitors within 4 weeks prior to study. Limited field external beam radiotherapy to prevent pathological fractures is allowed , when unirradiated, evaluable lesions elsewhere are present.
* Cardiac disease with New York Heart Association classification of III or IV
* Patients who are pregnant, nursing or of reproductive potential and are not practicing an effective method of contraception
* Any unrelated illness, e.g. active infection, inflammation, medical condition or laboratory abnormalities, which in the judgment of the investigator will significantly affect patients' clinical status
* Life expectancy shorter than 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Tumor response | 12 weeks
  Evaluation according to RECIST criteria

SECONDARY OUTCOMES:
Progression free survival | 3 years
  Progression free survival is defined as the time measured from the day of first administration of Lu-177-girentuximab to first progression or death, whichever comes first.
Toxicity | up to 14 weeks after last therapeutic infusion
  Toxicity defined by NCI Common Terminology Criteria for Adverse Events (CTCAE v3.0)

CONTACTS AND LOCATIONS:
Overall Officials: W. J. Oyen, MD, PhD, Principal Investigator — Department of Nuclear Medicine, Radboud University Medical Center Nijmegen; P. F. Mulders, MD, PhD, Principal Investigator — Department of Urology, Radboud University Medical Center Nijmegen
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Muselaers CH, Boers-Sonderen MJ, van Oostenbrugge TJ, Boerman OC, Desar IM, Stillebroer AB, Mulder SF, van Herpen CM, Langenhuijsen JF, Oosterwijk E, Oyen WJ, Mulders PF. Phase 2 Study of Lutetium 177-Labeled Anti-Carbonic Anhydrase IX Monoclonal Antibody Girentuximab in Patients with Advanced Renal Cell Carcinoma. Eur Urol. 2016 May;69(5):767-70. doi: 10.1016/j.eururo.2015.11.033. Epub 2015 Dec 23. PMID 26706103